CLINICAL TRIAL: NCT06695559
Title: Non Surgical Treatment of Peri-implantitis Using an Oscillating Chitosan Brush With Adjunctive Tetracycline Slurry: A Randomized Clinical Trial
Brief Title: Non-surgical Treatment of Peri-implantitis Using Chitosan Brush and Tetracycline Slurry
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200/16-06-2023
Record Dates: First submitted 2024-11-17; First posted 2024-11-19 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Periimplantitis; Periimplant Diseases
Keywords: non-surgical treatment; periimplantitis; chitosan; tetracycline
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Labrida Bioclean (Active Comparator): The implant pockets will be debrided with the Labrida BioClean™ biodegradable brush for 2 minutes and with the brush seated in an oscillating dental handpiece (NSK ESQ10 TEQ) and thereafter irrigated with sterile saline. The treatment will be repeated every three months. Debridement is performed with local anaesthesia as needed.
  Interventions: Other: Labrida Bioclean
- Labrida Bioclean and tetracycline slurry (Experimental): The implant pockets will be debrided with the BioClean™ biodegradable brush for 2 minutes and with the brush seated in an oscillating dental handpiece (NSK ESQ10 TEQ) and thereafter irrigated two minutes with tetracycline-hydrochloride (Arco Interpharma AS, Hokksund, Norway) in sterile saline with a concentration of 150 mg/ml, as chemical detergent adjunct to the chitosan brush. The treatment will be repeated every three months. Debridement is performed with local anaesthesia as needed.
  Interventions: Drug: Tetracycline slurry

INTERVENTIONS:
Other: Labrida Bioclean — Debridement on the active comparator group will be implemented on the implant surface with Labrida Bioclean (i.e. the chitosan brush).
  Arms: Labrida Bioclean
Drug: Tetracycline slurry — On the experimental group debridement of the implant surface will be carried out with Labrida Bioclean and thereafter irrigation of the periimplant sulcus with tetracycline slurry will take place.
  Other Names: Labrida Bioclean
  Arms: Labrida Bioclean and tetracycline slurry

SUMMARY:
Aim:

The aim of this prospective, randomized, parallel arm, blind clinical trial is to compare the clinical and radiographic outcomes following non-surgical treatment of mild peri-implant defects using Labrida Bioclean with or without the application of tetracycline slurry.

Research Hypothesis:

The hypothesis is that the adjunctive application of tetracycline slurry will enhance the clinical and radiographic results of non-surgical treatment of mild peri-implant defects (defined as peri-implant bone loss 3-6 mm with pocket depths 6 mm or deeper) with Labrida Bioclean. Probing pocket depth (PPD) reduction will be the primary outcome, whereas clinical attachment level (CAL), radiographic bone fill (RBF), recession depth (REC), modified bleeding index (mBI), presence of plaque (PL) , suppuration on probing (SUP) and Matrix Metalloproteinase-8 (MMP-8) levels on peri-implant sulcus fluid (PISF) will constitute the secondary outcome measures.

Groups:

Active comparator group: Debridement with Labrida Bioclean

Experimental group: Debridement with Labrida Bioclean and irrigation with tetracycline slurry

At the end of the treatment procedure patients will be given oral hygiene instructions and specifically patients of the experimental group will be instructed to refrain from oral hygiene for 24 hours before initiating oral hygiene. 1 month after therapy patients will be re-evaluated as a mean of PPD, CAL, REC, mBI, PL, SUP measurements and levels of MMP-8 on PISF. 3 months after therapy will be re-evaluated for second time as in the 1 month re-evaluation. Furthermore, treatment will be repeated as it was randomized on baseline. On 6 month re-evaluation PPD, CAL, REC, mBI, PL, SUP measurements will be made and also a periapical x-ray will be taken to compare the peri-implant bone level with the respective bone level on the x-ray of the baseline. On all of these appointments oral hygiene instructions and motivation will be given to the patients.

DETAILED DESCRIPTION:
Inflammation and loss of attachment around dental implants (i.e., peri-implantitis) is a growing issue within the field of dental implantology. Studies show that regular cleaning of dental implants is important to avoid progression of mucositis to peri-implantitis. Instruments specifically designed for this purpose are however scarce and mostly not scientifically validated with respect to efficacy and safety. Leaving remnants of the instrument on the implant surface or scratching the surface may also impede optimal peri-implant healing. Currently used maintenance procedures of implants comprise use of titanium curettes, plastic or carbon fiber curettes, ultrasound or lasers which is cumbersome, time consuming and in the example of lasers rather costly. Scientific evidence for the effectiveness of such interventions is also variable. It is also suggested that some procedures may even cause more problems rather than improving peri-implant health. One obvious risk factor is to leave foreign material, such as nylon, carbon or non-inert metals, in an environment comprising of bone, titanium implant and inflamed soft tissue which may cause a foreign body reaction and even further aggravation of the bone loss around the implant.

So far there is no device specifically developed for cleaning dental implants, neither with mucositis nor with mild peri-implantitis, and it is of utmost importance to develop methods optimized for therapy with the aim to prolong the life span of ailing dental implants.

As for the chitosan biodegradable brush, the brush bristles of the test device (BioClean Trademark - TM, LABRIDA AS, Oslo Norway) are made of the biopolymer chitosan. Any debris left from the chitosan bristles is completely biocompatible and will dissolve or be resorbed thus not causing harm to the tissues surrounding the implant. Chitosan is made from chitin derived from shell of marine crustaceans such as shrimp and crab, however chemically modified and thus not even considered to be animally derived. Chitosan has been approved for use in e.g., surgical bandages, as a haemostatic agent and as dietary supplement used in a wide range of nutritional and health products. Chitosan has also been documented to be non-allergenic and it has been suggested that chitosan has anti-inflammatory properties.

In three previous research project performed at the Department of Periodontology, Institute of Clinical Dentistry, University of Oslo the safety and potential to reduce peri-implant inflammation was tested. In the first study, which was a pilot consecutive case series of six months duration, 13 patients with 13 implants diagnosed with peri-implant mucositis were treated with the device. Significant improvements in parameters of inflammation were demonstrated up to 6 months after baseline treatment. In a randomized, split mouth, examiner blinded, clinical trial of 6 months duration, including 12 patients diagnosed with peri-implant mucositis the chitosan brush was compared with titanium curettes. Both groups demonstrated significant reductions in clinical parameters between baseline, 4 weeks and 6 months but the test implants treated with the chitosan brush had a better improvement in BoP (Bleeding on Probing) at 2 weeks and a better improvement in PPD (Probing Pocket Depth) at 2 weeks and 4 weeks as compared with the implants treated with the titanium curettes. None of the implants demonstrated progression in bone-loss during the course of the study. In recent multicenter consecutive case series in 6 centers in Sweden, Norway and Italy it was demonstrated that treatment with a chitosan brush of implants affected by mild peri-implantitis lead to a reduction in parameters of inflammation up to three months after baseline. No control group was however included in this study and it will be important to further evolve on these early results also comparing treatment with a chitosan brush with a more conventional treatment strategy.

Tetracycline has broad antimicrobial capabilities in addition to a low pH, which can aid in the cleaning of implant surfaces. Inhibition of collagenase is also an effect of localized applied tetracycline. In a recent study by Samuelsson, Valnes and Wohlfahrt 24 patients were treated with a protocol consisting of debridement with a chitosan brush seated in an oscillating dental handpiece with adjunct H2O2 3% and tetracycline slurry. In 21 patients with 23 implants, reductions in both the CAL and mBoP(modified Bleeding on Probing) were observed between baseline and the reexaminations between nine months and up to 43 months.

Developing simple non surgical protocols for treatment of peri-implantitis will have a tremendous value for patients to avoid high expenses and morbidity by avoiding surgical intervention

Aim:

The aim of this prospective, randomized, parallel arm, blind clinical trial is to compare the clinical and radiographic outcomes following non-surgical treatment of mild peri-implant defects using Labrida Bioclean with or without the application of tetracycline slurry.

Research Hypothesis:

The hypothesis is that the adjunctive application of tetracycline slurry will enhance the clinical and radiographic results of non-surgical treatment of mild peri-implant defects (defined as peri-implant bone loss 3-6 mm with pocket depths 6 mm or deeper, with mBI scores 2 or 3) with Labrida Bioclean. Probing pocket depth (PPD) reduction will be the primary outcome, whereas clinical attachment level (CAL), radiographic bone fill (RBF), recession depth (REC), modified bleeding index (mBI), presence of plaque (PL) , suppuration on probing (SUP) and MMP-8 levels on peri-implant sulcus fluid (PISF) will constitute the secondary outcome measures.

Study design:

The study will be a prospective, randomized, clinical trial of 6 months duration.

Treatment allocation:

Patients will be allocated either to test (BioClean with tetracycline slurry) or control (BioClean alone) treatment by computer-generated block randomization to ensure equal sample sizes. A software (www.randomizer.org) will be used by one of the investigators who will not participate in the clinical and radiographic measurements nor the therapeutic intervention, to generate a block randomization. Thus, participants will be randomized in one of the two groups. In patients with more than one implant meeting the inclusion criteria, a second randomization scheme with the same software will take place, to determine which will be included. The randomization results will be placed in sealed envelopes accessible only to the principal investigator and opened for each patient after the end of debridement with Labrida Bioclean to determine if tetracycline slurry will be applied or not Study setting Patient screening, inclusions and all clinical examinations will be performed by a board-certified specialist in periodontology or by a post-graduate student of the department of Preventive Dentistry, Periodontology & Implant Biology. Treatments will be performed by a board-certified specialist in periodontology or by a post-graduate student of the department of Preventive Dentistry, Periodontology & Implant Biology.

Patients:

40 patients (20+20) diagnosed with mild peri-implantitis, defined as peri-implant bone loss 3 -6 mm (minimum 3 mm and maximum 6 mm) with PPD 6 mm or deeper with mBI scores 2 or 3, will be included.

Recruitment of patients:

Patients referred to the specialist clinic in periodontology, will be screened for inclusion.

Procedure:

Before initiation of the study, the protocol will be approved by the Ethics Committee of the Dental School of the Aristotle University of Thessaloniki. In addition, informed consent will be signed by all participants.

Prior to inclusion in the study, an initial examination will be performed, including medical history, full- mouth plaque and bleeding scores, and PPDs, CALs, RECs, SUP, mBI, PL at 6 points on each implant. In addition, oral hygiene instructions and motivation will be given. Patients will receive a supragingival debridement with ultrasonic instruments, in one session, without local anesthesia. Commercially available and specific for implant debridement titanium curettes will be used to remove any supramucosal calculus in both groups prior to test or control treatments. Patients diagnosed with periodontal disease should be in the state of reminiscence after finished and re-evaluated active periodontal therapy. Endodontic lesions and dental decay should be treated prior to study start. Plaque Index (dichotomous scoring) should be below 20%. Before the treatment PISF sample will be collected for evaluation of MMP-8 levels with ELISA.

Active comparator group: Debridement with Labrida Bioclean Experimental group: Debridement with Labrida Bioclean and irrigation with tetracycline slurry

Treatment procedures:

Active comparator group: The implant pockets will be debrided with the Labrida BioClean biodegradable brush for 2 minutes and with the brush seated in an oscillating dental handpiece (NSK ESQ10 TEQ) and thereafter irrigated with sterile saline. The treatment will be repeated every three months. Debridement is performed with local anaesthesia as needed.

Experimental group: The implant pockets will be debrided with the BioClean biodegradable brush for 2 minutes and with the brush seated in an oscillating dental handpiece (NSK ESQ10 TEQ) and thereafter irrigated two minutes with tetracycline-hydrochloride (Arco Interpharma AS, Hokksund, Norway) in sterile saline with a concentration of 150 mg/ml, as chemical detergent adjunct to the chitosan brush. The treatment will be repeated every three months. Debridement is performed with local anaesthesia as needed.

At the end of the treatment procedure patients will be given oral hygiene instructions and specifically patients of the experimental group will be instructed to refrain from oral hygiene for 24 hours before initiating oral hygiene. 1 month after therapy patients will be re-evaluated as means of PPD, CAL, REC, mBI, PL, SUP measurements and levels of MMP-8 on PISF. 3 months after therapy will be re-evaluated for second time as in the 1 month re-evaluation. Furthermore, treatment will be repeated as it was randomized on baseline. On 6 month re-evaluation PPD, CAL, REC, mBI, PL, SUP measurements will be made and also a periapical x-ray will be taken to compare the peri-implant bone level with the respective bone level on the x-ray of the baseline. On all of these appointments oral hygiene instructions and motivation will be given to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Peri-implantitis defined as periimplant bone loss ≥ 3 mm on periapical x-rays distally, mesially or both and with Probing Pocket Depth (PPD) ≥6 mm.
* Peri-implantitis as defined above on an implant that has been in function for more than 12 months prior to study start.
* Above 18 years of age.
* Eligible for treatment in an outpatient dental clinic (ie, American Society of Anesthesiologists classification I and II).
* Had full-mouth plaque scores < 20% prior to final inclusion.
* Had at least one implant with a loading time of ≥ 12 months prior to baseline.
* Signed Informed Consent obtained prior to start.
* Psychological appropriateness
* Consent to complete all follow-up visits.
* Patients diagnosed with periodontal disease must have undergone causative treatment and be re-evaluated

Exclusion Criteria:

* Peri-implant bone loss > 6 mm on periapical x-rays
* Cemented supraconstructions and/or screw retained supraconstructions that for technical reasons makes it impossible to access implant for clinical measurements.
* Technical complications which according to the examiners judgement has contributed to the disease state and not possible to resolve prior to final inclusion.
* Mobile implant.
* Implants previously treated for peri-implantitis with grafting materials.
* Receiving medications known to induce mucosal hyperplasia.
* Uncontrolled diabetes (HbA1c > 7).
* Receiving systemic antibiotics < 3 months prior to inclusion.
* Pregnant or lactating.
* Any condition or current treatment for any condition, which in the opinion of the investigator and/or consulting physician, may constitute an unwarranted risk.
* Presence of psychological characteristics, such as inappropriate attitude or motivation, which will influence treatment execution and treatment outcome.
* Unwillingness to undergo treatment.
* If, in the medical opinion of the therapist, conditions are such that dental implants are deemed failing.
* Ongoing or previous radiotherapy to the head-neck region.
* Ongoing or previous chemotherapy.
* Systemic long-term corticosteroid treatment.
* Patients medicating with warfarin products or similar

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth | Change from baseline to 6 months
  Pocket depth of periimplant sulcus measured in millimeters

SECONDARY OUTCOMES:
Radiographic bone fill | Change from baseline to 6 months
  Bone level of the periimplant defect
Clinical attachment level | Change from baseline to 6 months
  Clinical attachment level measured in millimeters
Recession | Change from baseline to 6 months
  Recession depth calculated as the difference of clinical attachment level minus probing depth
Presence of plaque | Change from baseline to 6 months
  Presence or absence of plaque (dichotomous scoring)
Modified Bleeding Index | Change from baseline to 6 months
  0: no bleeding, 1: isolated bleeding spots visible, 2: blood forms a confluent red line on margin, 3: heavy or profuse bleeding
MMP-8 levels | Change from baseline to 3 months
  Levels of MMP-8 on periimplant sulcus fluid that will be analyzed with ELISA
Suppuration on probing | Change from baseline to 6 months
  Presence or absence of suppuration within 30 seconds following probing of the pocket (dichotomous scoring)

CONTACTS AND LOCATIONS:
Overall Officials: Lazaros Tsalikis, Study Director — Professor
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koldsland OC, Scheie AA, Aass AM. Prevalence of peri-implantitis related to severity of the disease with different degrees of bone loss. J Periodontol. 2010 Feb;81(2):231-8. doi: 10.1902/jop.2009.090269. PMID 20151801
- [Background] Costa FO, Takenaka-Martinez S, Cota LO, Ferreira SD, Silva GL, Costa JE. Peri-implant disease in subjects with and without preventive maintenance: a 5-year follow-up. J Clin Periodontol. 2012 Feb;39(2):173-81. doi: 10.1111/j.1600-051X.2011.01819.x. Epub 2011 Nov 23. PMID 22111654
- [Background] Sorsa T, Ding Y, Salo T, Lauhio A, Teronen O, Ingman T, Ohtani H, Andoh N, Takeha S, Konttinen YT. Effects of tetracyclines on neutrophil, gingival, and salivary collagenases. A functional and western-blot assessment with special reference to their cellular sources in periodontal diseases. Ann N Y Acad Sci. 1994 Sep 6;732:112-31. doi: 10.1111/j.1749-6632.1994.tb24729.x. PMID 7978785
- [Background] Mensi M, Scotti E, Calza S, Pilloni A, Grusovin MG, Mongardini C. A new multiple anti-infective non-surgical therapy in the treatment of peri-implantitis: a case series. Minerva Stomatol. 2017 Dec;66(6):255-266. doi: 10.23736/S0026-4970.17.04054-7. Epub 2017 Oct 3. PMID 28975771
- [Background] Mombelli A, Feloutzis A, Bragger U, Lang NP. Treatment of peri-implantitis by local delivery of tetracycline. Clinical, microbiological and radiological results. Clin Oral Implants Res. 2001 Aug;12(4):287-94. doi: 10.1034/j.1600-0501.2001.012004287.x. English, French, German. PMID 11488856
- [Background] Roos-Jansaker AM, Renvert H, Lindahl C, Renvert S. Submerged healing following surgical treatment of peri-implantitis: a case series. J Clin Periodontol. 2007 Aug;34(8):723-7. doi: 10.1111/j.1600-051X.2007.01098.x. Epub 2007 May 29. PMID 17535286
- [Background] Samuelsson RS, Valnes AK, Wohlfahrt JC. Nonsurgical Treatment of Peri-implantitis Using a Chitosan Brush with Adjunctive Chemical Decontaminants- A Retrospective Case Series. Int J Oral Maxillofac Implants. 2022 Nov-Dec;37(6):1261-1267. doi: 10.11607/jomi.9602. PMID 36450034
- [Background] Khan SN, Koldsland OC, Roos-Jansaker AM, Wohlfahrt JC, Verket A, Mdala I, Magnusson A, Salvesen E, Hjortsjo C. Non-surgical treatment of mild to moderate peri-implantitis using an oscillating chitosan brush or a titanium curette-A randomized multicentre controlled clinical trial. Clin Oral Implants Res. 2022 Dec;33(12):1254-1264. doi: 10.1111/clr.14007. Epub 2022 Oct 18. PMID 36207993
- [Background] Wohlfahrt JC, Evensen BJ, Zeza B, Jansson H, Pilloni A, Roos-Jansaker AM, Di Tanna GL, Aass AM, Klepp M, Koldsland OC. A novel non-surgical method for mild peri-implantitis- a multicenter consecutive case series. Int J Implant Dent. 2017 Dec;3(1):38. doi: 10.1186/s40729-017-0098-y. Epub 2017 Aug 3. PMID 28776288